CLINICAL TRIAL: NCT05461157
Title: The Application of Preoperative Silicone Ointment and Its Effect on Wound Healing
Brief Title: Preoperative Silicone Ointment and Wound Healing
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Biodermis (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2000033013_a
Record Dates: First submitted 2022-07-06; First posted 2022-07-15 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Wound Heal; Scar; Scar, Hypertrophic; Keloid; Keloid Scar Following Surgery; Surgical Incision
Keywords: Wound healing; Surgical incision; Scar; Hypertrophic scar; Keloid; Silicone ointment
MeSH Terms: conditions — Cicatrix; Cicatrix, Hypertrophic; Keloid; Surgical Wound

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either silicone ointment or placebo ointment prior to undergoing scheduled surgery. After surgery, all participants will use silicone ointment.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Preoperative silicone ointment (Experimental): Participants will apply silicone ointment to the area where the surgical incision will be made, twice daily for 2-6 weeks prior to their scheduled surgery.
  Interventions: Device: Preoperative silicone ointment
- Preoperative placebo ointment (Placebo Comparator): Participants will apply placebo ointment to the area where the surgical incision will be made, twice daily for 2-6 weeks prior to their scheduled surgery.
  Interventions: Other: Preoperative placebo ointment

INTERVENTIONS:
Device: Preoperative silicone ointment — The silicone ointment in this study is the Biodermis Scar Aid Silicone Stick, an FDA-approved silicone ointment that is available for purchase over the counter.
  Other Names: Biodermis Scar Aid Silicone Stick
  Arms: Preoperative silicone ointment
Other: Preoperative placebo ointment — The placebo ointment in this study is a generic, non-flavored lip balm that is identical in packaging and texture to the Biodermis Scar Aid Silicone Stick used in the treatment arm.
  Other Names: Lip balm
  Arms: Preoperative placebo ointment

SUMMARY:
Optimal scar healing is of great importance to patients, especially following surgery of the head and neck. This study evaluates the effectiveness of preoperative silicone ointment in wound healing in head and neck surgeries.

DETAILED DESCRIPTION:
Following surgical procedures, the formation of hypertrophic scars and keloids affects patients' well-being, including quality of life and mental/psychological health. Scars in certain areas, including the face, neck, ears, and upper chest and back, are especially likely to develop abnormally. Due to these adverse outcomes, patients often request products and procedures that will improve the appearance of scars. Few studies have addressed preoperative measures that can improve scar healing.

Surgeons often recommend that patients apply moisturizing ointments to the area of the incision prior to surgery; however, this is based on clinical consensus and is not evidence-based. Silicone products are understood to promote hydration of the skin and are considered first-line prophylactic and treatment therapy for abnormal scars (hypertrophic scars and keloids) when used after a surgery or injury. This study seeks to evaluate preoperative application of silicone ointment and its effect on surgical scar healing.

The success of surgical scar healing will be determined by researcher and participant ratings on validated scar assessment scales. The secondary objective of this study is to evaluate the effect of preoperative application of silicone ointment on postoperative wound complications.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo non-emergent surgery of the head and/or neck for a benign (non-cancerous) condition
* Able to comply with all study procedures for the duration of the study
* Provision of signed and dated informed consent form

Exclusion Criteria:

* Current use of products intended to improve scar healing (silicone or otherwise); skincare products not specifically marketed for scar healing are acceptable
* Known allergic reactions to components of the silicone ointment
* Dermatologic conditions that disrupt the integrity of the skin, e.g. severe acne, psoriasis
* Need for tracheostomy postoperatively
* Have any form of active malignancy at the time of surgery
* Have a history of radiation involving the surgical site
* Prior surgery involving all or part of the planned surgical incision
* Current use of chronic steroids or other immunosuppressive medications
* Lack of decision-making capacity
* Not fluent in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-11-14 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Short-term wound healing measured by the Patient and Observer Scar Assessment Scale (POSAS) | 3 months after surgery
  The Patient and Observer Scar Assessment Scale (POSAS) includes two components: an observer's evaluation of a scar and a patient's evaluation of a scar. The Patient Scar Assessment Scale component asks the patient the degree to which the scar is painful or itchy, how the color, stiffness, thickness, and irregularity of the scar compare to the patient's normal skin, and the patient's overall opinion of the scar. Each question is scored on a scale of 1 (not at all painful, itchy, or different) to 10 (very much painful, itchy, or different), and the numbers are totaled to produce a final score. The Observer Scar Assessment Scale component measures vascularity, pigmentation, thickness, relief, pliability, and surface area, as well as the observer's overall opinion of the scar. Each question is scored on a scale of 1 (like normal skin) to 10 (worst scar imaginable), and the numbers are totaled to produce a final score.
Long-term wound healing measured by the Patient and Observer Scar Assessment Scale (POSAS) | 12 months after surgery
  The Patient and Observer Scar Assessment Scale (POSAS) includes two components: an observer's evaluation of a scar and a patient's evaluation of a scar. The Patient Scar Assessment Scale component asks the patient the degree to which the scar is painful or itchy, how the color, stiffness, thickness, and irregularity of the scar compare to the patient's normal skin, and the patient's overall opinion of the scar. Each question is scored on a scale of 1 (not at all painful, itchy, or different) to 10 (very much painful, itchy, or different), and the numbers are totaled to produce a final score. The Observer Scar Assessment Scale component measures vascularity, pigmentation, thickness, relief, pliability, and surface area, as well as the observer's overall opinion of the scar. Each question is scored on a scale of 1 (like normal skin) to 10 (worst scar imaginable), and the numbers are totaled to produce a final score.
Short-term wound healing measured by the Scar Cosmesis Assessment and Rating (SCAR) Scale | 3 months after surgery
  The Scar Cosmesis Assessment and Rating (SCAR) scale is a validated measure consisting of both observer and patient evaluations. The observer assesses scar spread, erythema, dyspigmentation, suture marks, hypertrophy or atrophy, and overall impression. The patient reports whether the scar is itchy or painful. The SCAR scale can be used to assess scars in person or photos of scars. The total possible score ranges from 0 (best possible scar) to 15 (worst possible scar).
Long-term wound healing measured by the Scar Cosmesis Assessment and Rating (SCAR) Scale | 12 months after surgery
  The Scar Cosmesis Assessment and Rating (SCAR) scale is a validated measure consisting of both observer and patient evaluations. The observer assesses scar spread, erythema, dyspigmentation, suture marks, hypertrophy or atrophy, and overall impression. The patient reports whether the scar is itchy or painful. The SCAR scale can be used to assess scars in person or photos of scars. The total possible score ranges from 0 (best possible scar) to 15 (worst possible scar).

SECONDARY OUTCOMES:
Length of hospital stay | 30 days after surgery
  Number of days a participant stays in the hospital following their scheduled surgery
Discharge location | 30 days after surgery
  Location (e.g. home, skilled nursing facility, etc.) to which a participant is discharged following surgery
Number of readmissions | 1 year after surgery
  Number of times a participant is readmitted to the hospital
Need for follow-up | 1 year after surgery
  Number of clinic or emergency department (ED) visits that are not part of the participant's routine care
Wound complications | 1 year after surgery
  Whether the participant had unexpected complications including infection, excessive bleeding, or dehiscence

CONTACTS AND LOCATIONS:
Overall Officials: Yan Lee, MD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] O'Brien L, Jones DJ. Silicone gel sheeting for preventing and treating hypertrophic and keloid scars. Cochrane Database Syst Rev. 2013 Sep 12;2013(9):CD003826. doi: 10.1002/14651858.CD003826.pub3. PMID 24030657
- [Background] Tran B, Wu JJ, Ratner D, Han G. Topical Scar Treatment Products for Wounds: A Systematic Review. Dermatol Surg. 2020 Dec;46(12):1564-1571. doi: 10.1097/DSS.0000000000002712. PMID 32932267
- [Background] Balci DD, Inandi T, Dogramaci CA, Celik E. DLQI scores in patients with keloids and hypertrophic scars: a prospective case control study. J Dtsch Dermatol Ges. 2009 Aug;7(8):688-92. doi: 10.1111/j.1610-0387.2009.07034.x. Epub 2009 Feb 18. English, German. PMID 19243478